CLINICAL TRIAL: NCT02427217
Title: A Multicenter Study on the Retrospective Safety and Efficacy of Fibrinogen Concentrate (Human) (FCH) for Routine Prophylaxis, Treatment of Bleeding or Surgery in Subjects With Congenital Fibrinogen Deficiency With a Prospective Followup Component
Brief Title: An Observational Cohort Study of the Safety and Efficacy of Fibrinogen Concentrate, Human (FCH) in Subjects With Congenital Fibrinogen Deficiency
Status: Completed | Type: Observational
Sponsor: CSL Behring (Industry)
Responsible Party: Sponsor
Other Study IDs: BI3023_4003
Record Dates: First submitted 2015-04-22; First posted 2015-04-27 (Estimated); Last update posted 2018-01-17 (Actual); Status verified 2018-01

CONDITIONS: Congenital Fibrinogen Deficiency
MeSH Terms: interventions — Fibrinogen

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other

GROUPS / COHORTS (1):
- Fibrinogen Concentrate, Human (FCH): A cohort of subjects who have retrospectively received FCH for the treatment of bleeding, routine prophylaxis and/or use in surgery, and who may continue to prospectively receive FCH at the discretion of the treating physician.
  Interventions: Biological: FCH

INTERVENTIONS:
Biological: FCH — FCH is a heat-treated, lyophilized fibrinogen (coagulation factor I) powder made from pooled human plasma. FCH is administered as an IV infusion.
  Other Names: Haemocomplettan® P; RiaSTAP®

SUMMARY:
This is a multicenter, non interventional, retrospective cohort study with a prospective, observational follow-up component to investigate the safety and efficacy of FCH use in subjects with congenital fibrinogen deficiency. Data will be collected on the safety and efficacy of FCH as used for the treatment of acute bleeding episodes, routine prophylaxis and perioperative bleeding in these subjects. All subjects have received FCH and may continue to receive FCH at the discretion of the treating physician / Primary Investigator according to the standard of care at the participating study site.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects of any age with a diagnosis of congenital fibrinogen deficiency.
* Have received FCH (Haemocomplettan® P or RiaSTAP®) for treatment of bleeding, surgery or prophylaxis.

Exclusion Criteria:

None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A cohort of subjects who have retrospectively received FCH for the treatment of bleeding, routine prophylaxis and/or use in surgery, and who may continue to prospectively receive FCH at the discretion of the treating physician.
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2015-05-07 (Actual); Primary Completion 2017-12-06 (Actual); Study Completion 2017-12-06 (Actual)

PRIMARY OUTCOMES:
Percentage of participants achieving hemostatic efficacy - retrospective | From the subject's first use of FCH, up to approximately 20 years.
  The investigator's overall assessment of hemostatic efficacy of FCH from a review of the subject's historical records.

SECONDARY OUTCOMES:
Percentage of participants achieving hemostatic efficacy - prospective | Approximately 12 months
  The investigator's overall assessment of hemostatic efficacy of FCH during the prospective follow-up period.
Percentage of participants with adverse events | Retrospective data collection is from the subject's first use of FCH (up to approximately 20 years); Prospective data collection is from the time of informed consent up to approximately 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Program Director, Study Director — CSL Behring
Locations (10):
- United States (3):
  - Study Site, Aurora, Colorado
  - Study Site, Las Vegas, Nevada
  - Study Site, Durham, North Carolina
- Canada (7):
  - Study Site, Calgary, Alberta
  - Study Site, Edmonton, Alberta
  - Study Site, Winnipeg, Manitoba
  - Study Site, Halifax, Nova Scotia
  - Study Site, Hamilton, Ontario
  - Study Site, Toronto, Ontario
  - Study Site, Montreal, Quebec